CLINICAL TRIAL: NCT03550391
Title: A Phase III Trial of Stereotactic Radiosurgery Compared With Hippocampal-Avoidant Whole Brain Radiotherapy (HA-WBRT) Plus Memantine for 5 or More Brain Metastases
Brief Title: Stereotactic Radiosurgery Compared With Hippocampal-Avoidant Whole Brain Radiotherapy (HA-WBRT) Plus Memantine for 5 or More Brain Metastases
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: Alliance for Clinical Trials in Oncology (Other); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCTG CE.7; NCI-2018-00395 (Other: NCI CTRP)
Record Dates: First submitted 2018-04-30; First posted 2018-06-08 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-04

CONDITIONS: Brain Metastases
MeSH Terms: conditions — Brain Neoplasms | interventions — Memantine; Radiotherapy; Radiosurgery

STUDY DESIGN:
Intervention Model Description: This is an international multi-centre, open-label, randomized phase III trial comparing stereotactic radiosurgery compared with hippocampal-avoidant whole brain radiotherapy (HA-WBRT) plus memantine for 5-15 brain metastases
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Hippocampal-avoidant (HA-WBRT) plus Memantine (Experimental): WBRT 30Gy in 10 fractions + memantine
  Interventions: Drug: Memantine; Radiation: Hippocampal-avoidant (HA-WBRT) Radiotherapy
- Stereotactic Radiosurgery (SRS) (Experimental): SRS 18-20 or 22Gy in single fraction
  Interventions: Procedure: Stereotactic Radiosurgery (SRS)

INTERVENTIONS:
Drug: Memantine — 20 mg (10 mg divided twice daily). Dose will be escalated by 5 mg per week. Memantine should start at 5 mg, and then increased in 5 mg increments at the following schedule, depending on the patient's response and tolerance:
  Arms: Hippocampal-avoidant (HA-WBRT) plus Memantine
Radiation: Hippocampal-avoidant (HA-WBRT) Radiotherapy — 30Gy in 10 fractions
  Arms: Hippocampal-avoidant (HA-WBRT) plus Memantine
Procedure: Stereotactic Radiosurgery (SRS) — 18-20 or 22 Gy in single fraction
  Arms: Stereotactic Radiosurgery (SRS)

SUMMARY:
Stereotactic radiosurgery (SRS) is a commonly used treatment for brain tumors. It is a one-day (or in some cases two day), out-patient procedure during which a high dose of radiation is delivered to small spots in the brain while excluding the surrounding normal brain.

Whole brain radiation therapy with hippocampal avoidance (HA-WBRT) is when radiation therapy is given to the whole brain, while trying to decrease the amount of radiation that is delivered to the area of the hippocampus. The hippocampus is a brain structure that is important for memory. Memantine is a drug that is given to help relieve symptoms that can be caused by WBRT, including problems with memory and other mental symptoms.

Health Canada, the regulatory body that oversees the use of drugs in Canada, has not approved the sale or use of memantine in combination with WBRT to treat this kind of cancer, although they have allowed its use in this study.

DETAILED DESCRIPTION:
The purpose of this research study is to compare the effects (good or bad) of receiving stereotactic radiosurgery (SRS) versus receiving hippocampal-avoidant whole brain radiotherapy (HA-WBRT) plus a drug called memantine, on brain metastases. Receiving SRS could control cancer that has spread to the brain.

This study will allow the researchers to know whether this different approach is better, the same, or worse than the usual approach. To decide if it is better, the study doctors will be looking to see if the stereotactic radiosurgery (SRS) helps to either slow the growth of cancer or stop it from coming back, compared to the usual approach. Doctors will also look to see if this new approach increases the life span of patients with this type of cancer, and if it helps with quality of life and cancer related symptoms.

The usual approach for patients who are not in a study is treatment with whole brain radiation therapy alone (WBRT).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have 5 or more brain metastases as counted on a T1 contrast enhanced MRI obtained ≤ 30 days from randomization (maximum 15 brain metastases).
* Patients must have a pathological diagnosis (cytological or histological) of a non-hematopoietic malignancy.
* The largest brain metastasis must measure <2.5 cm in maximal diameter.
* Centre must have the ability to treat patients with either a Gamma Knife, Cyberknife, or a linear accelerator-based radiosurgery system.
* Patient must be > 18 years of age.
* Patient is able (i.e. sufficiently fluent) and willing to complete the quality of life questionnaires in either English or French either alone or with assistance.
* ECOG performance status 0, 1, or 2.
* Creatinine clearance must be ≥ 30 ml/min within 28 days prior to registration.
* The Neurocognitive Testing examiner must have credentialing confirming completion of the neurocognitive testing training.
* Facility is credentialed by IROC to perform SRS and HA-WBRT. The treating centre must have completed stereotactic radiosurgery credentialing of the specific system(s) to be used in study patients. The treating centre must have completed IMRT credintialing of this specific IMRT systems to be used in study patients for the purposes of HA-WBRT.
* Patient consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each patient must sign a consent form prior to enrolment in the trial to document their willingness to participate.
* A similar process must be followed for sites outside of Canada as per their respective cooperative group's procedures.
* Patients must be accessible for treatment and follow-up. Investigators must assure themselves the patients randomized on this trial will be available for complete documentation of the treatment, adverse events, and follow-up.
* In accordance with CCTG policy, protocol treatment is to begin within 14 days of patient enrolment.
* Women/men of childbearing potential must have agreed to use a highly effective contraceptive method.

Exclusion Criteria:

* Pregnant or nursing women.
* Men or women of childbearing potential who are unwilling to employ adequate contraception.
* Inability to complete a brain MRI.
* Known allergy to gadolinium.
* Prior cranial radiation therapy.
* Planned cytotoxic chemotherapy within 48 hours prior or after the SRS or HA-WBRT.
* Primary germ cell tumour, small cell carcinoma, or lymphoma.
* Widespread definitive leptomeningeal metastasis. This includes cranial nerve palsy, leptomeningeal carcinomatosis, ependymal involvement, cranial nerve involvement on imaging, suspicious linear meningeal enhancement, or cerebrospinal fluid (CSF) positive for tumour cells.
* A brain metastasis that is located ≤ 5 mm of the optic chiasm or either optic nerve.
* Surgical resection of a brain metastasis (stereotactic biopsies will be allowed).
* More than 15 brain metastases on a volumetric T1 contrast MRI (voxels of 1mm or smaller) performed within the past 14 days, or more than 10 metastases in the case of a non-volumetric MRI.
* Prior allergic reaction to memantine.
* Current alcohol or drug abuse.
* Current use of NMDA antagonists, such as amantadine, ketamine, or dextromethorphan.
* Diagnosis of chronic liver disease/cirrhosis of the liver (e.g. Child-Pugh class B or C).
* Patients with architectural distortion of lateral ventricular systems, which, in the opinion of the local investigator, makes hippocampal delineation challenging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2018-11-22 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 4.5 years
  To compare the overall survival in patients with five to fifteen brain metastases who receive SRS compared to patients who receive HA-WBRT + memantine
Neurocognitive progression-free survival | 4.5 years
  To compare the neurocognitive progression-free survival in patients with five to fifteen brain metastases who receive SRS compared to patients who receive HA-WBRT + memantine

SECONDARY OUTCOMES:
Time to central nervous system (CNS) failure (local, distant, and leptomeningeal) in patients who receive SRS compared to patients who receive HA-WBRT + memantine | 4.5 years
Difference in CNS failure patterns (local, distant, or leptomeningeal) in patients who receive SRS compared to patients who receive HA-WBRT + memantine | 4.5 years
Number of salvage procedures following SRS in comparison to HA-WBRT + memantine | 4.5 years
Neurocognitive progression-free survival in patients who receive SRS compared to HA-WBRT + memantine | 4.5 years
  measured from date the patient is randomized to date at which there is a drop of at least 1.5 standard deviations from baseline in two of the six neurocognitive tests (all tests are standardized based on published norms)
Tabulate and descriptively compare the post-treatment adverse events associated with the interventions. | 4.5 years
Time delay to (re-)initiation of systemic therapy in patients receiving SRS in comparison to HA-WBRT + memantine | 4.5 years
Prospectively validate a predictive nomogram for distant brain failure in patients who receive SRS | 4.5 years
  a predictive nomogram as a clinically useful tool to determine the likelihood of distant brain failure (DBF) at different time points after radiosurgery
Compare the estimated cost of brain-related therapies in patients who receive SRS compared to patients who receive HA-WBRT + memantine. | 4.5 years
  Comparison based on payer rates (Medicare for US / provincial heath authorities in Canadian jurisdictions with activity-based funding)
Quality of life, as assessed by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (QLQ-C30) with brain cancer module (BN20) | 4.5 years
Quality of life assessed by ECOG performance status | 4.5 years
Quality of life, as assessed by EQ-5D-5L | 4.5 years
Collect plasma to evaluate whether detectable somatic mutations in liquid biopsy can enhance prediction of the overall survival and development of new brain metastases. | 4.5 years
Analysis of serum samples for inflammatory biomarker C-reactive protein and brain-derived-neurotrophic factor (BDNF) to elucidate molecular/genomic mechanisms of neurocognitive decline and associated radiographic changes | 4.5 years
Collect whole-brain dosimetry in SRS patients to be prospectively correlated with cognitive toxicity, intracranial control and radiation necrosis | 4.5 years
Evaluate serial changes in imaging features found in routine MRI images (T2w changes, morphometry) that may predict tumour control and/or neurocognitive outcomes | 4.5 years

CONTACTS AND LOCATIONS:
Overall Officials: David Roberge, Study Chair — CHUM-Centre Hospitalier de l'Universite de Montreal; Michael Chan, Study Chair — Wake Forest School of Medicine, Winston-Salem, NC; Vina Gondi, Study Chair — Northwestern Medicine Cancer Center, Warrenville IL
Locations (86):
- United States (73):
  - University of Arizona Cancer Center-Orange Grove Campus, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - City of Hope Corona, Corona, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - City of Hope at Irvine Lennar, Irvine, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - City of Hope Antelope Valley, Lancaster, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Kaiser Permanente-Rancho Cordova Cancer Center, Rancho Cordova, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - South Sacramento Cancer Center, Sacramento, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - City of Hope South Pasadena, South Pasadena, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - City of Hope South Bay, Torrance, California
  - City of Hope Upland, Upland, California
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Memorial Hospital West, Pembroke Pines, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Northwestern University, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - HSHS Saint Elizabeth's Hospital, O'Fallon, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Community Cancer Center North, Indianapolis, Indiana
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Luminis Health Anne Arundel Medical Center, Annapolis, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - AtlantiCare Surgery Center, Egg Harbor, New Jersey
  - State University of New York Upstate Medical University, Syracuse, New York
  - SUNY Upstate Medical Center-Community Campus, Syracuse, New York
  - Mission Hospital, Asheville, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Fox Chase Cancer Center Buckingham, Furlong, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Self Regional Healthcare, Greenwood, South Carolina
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Dartmouth Cancer Center - North, Saint Johnsbury, Vermont
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (13):
  - Arthur J E Child Comprehensive Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - QEII Health Sciences Centre/Nova Scotia Health Authority, Halifax, Nova Scotia
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - London Regional Cancer Program, London, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - CSSS Champlain-Charles Le Moyne, Greenfield Park, Quebec
  - CHUM - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - The Research Institute of the McGill University Health Centre (MUHC), Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - CHU de Quebec-L'Hotel-Dieu de Quebec (HDQ), Québec, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke-Fleurimont, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No